CLINICAL TRIAL: NCT05133401
Title: The Role of Imaging Techniques in Predicting Double-Lumen Tube Size and Positioning. Prospective Observational Study.
Brief Title: Can Imaging Techniques Contribute to the Proper Insertion of Double-lumen Tubes?
Status: Completed | Type: Observational
Sponsor: Atatürk Chest Diseases and Chest Surgery Training and Research Hospital (Other)
Responsible Party: Principal Investigator, Ali Alagoz, Principal Investigator, Atatürk Chest Diseases and Chest Surgery Training and Research Hospital
Other Study IDs: 2012-KAEK-15/2231
Record Dates: First submitted 2021-11-04; First posted 2021-11-24 (Actual); Last update posted 2022-01-24 (Actual); Status verified 2022-01

CONDITIONS: Double-Lumen Tube; Ultrasonography; Computed Tomography

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: Ultrasound-guided tracheal width measurement — Ultrasound measurements will be made with a 5-10 MegaHertz linear probe positioned in the horizontal plane at the midline of the anterior neck. After identifying the vocal cords as paired hyperechoic linear structures, the probe was moved caudally to visualize the cricoid arch. The transverse air column diameter was measured at the lower border of the cricoid cartilage.

SUMMARY:
In thoracic surgery, one-lung ventilation using a double-lumen tube (DLT) is often performed to protect dependent lung and provide comfortable surgical conditions. However, serious complications and adverse events can be encountered during DLT placement. One of the most important steps to avoid these drawbacks is to choose the appropriate size of DLT. The width of the trachea can be measured by using different imaging methods such as computed tomography (CT) and ultrasonography (US) to predict the appropriate DLT size. CT can also contribute to the proper placement of DLT by giving us the length of the trachea and main bronchi. In this study, we hypothesized that the size of the DLT can be determined more accurately by measuring the trachea diameter by using US and CT before DLT intubation. At the same time, we aimed to determine whether the evaluation of tracheobronchial anatomy with CT would contribute to the placement of DLT at a more appropriate level.

ELIGIBILITY:
Inclusion Criteria:

* Patients who will undergo elective thoracotomy or video-assisted thoracic surgery with general anesthesia with DLT intubation
* BMI 18 - 35 kg/m2
* Age 18 - 80 years old

Exclusion Criteria:

* Mallampati score 3 and 4
* History of tracheostomy, tracheal deviation, or distortion
* Emergency surgery

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: A total of 100 patients with a body mass index between18-35 kg/m2 in the ASA I-II-III risk group, aged 18-80, who will undergo elective thoracic surgery, require intubation with a double-lumen tube will be included in the study.
Sampling Method: Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2021-06-01 (Actual); Primary Completion 2021-11-30 (Actual); Study Completion 2021-12-30 (Actual)

PRIMARY OUTCOMES:
The measurement of the trachea diameter with ultrasound determines the size of the double-lumen tube to be used. | 1 hour
  After measuring the diameter of the trachea with ultrasound, the doctor will determine the double-lumen tube to be used according to the ultrasound measurement. Another experienced anesthesiologist, unaware of this result, will insert the double-lumen tube that he has determined with the conventional method.
The measurement of the trachea diameter by computerized tomography determines the size of the double-lumen tube is used. | 1 hour
  After measuring the diameter of the trachea with computerized tomography, the doctor will determine the double-lumen tube to be used according to the computerized tomography measurement. Another experienced anesthesiologist, unaware of this result, will insert the double-lumen tube that he has determined with the conventional method.
The measurement of the tracheal and main bronchi length and main bronchi diameter by computerized tomography in determining the size of the double-lumen tube and proper positioning of the double-lumen tube. | 1 hour
  The correlation of predicted and used DLT size. In addition, the correlation between DLT malposition rate and trachea and main bronchi length and main bronchi diameter measured by imaging methods.

SECONDARY OUTCOMES:
Complications related to double-lumen tube intubation | 1 day
  Evaluation of trauma, bleeding, sore throat and hoarseness in the airways due to double-lumen tube intubation.

CONTACTS AND LOCATIONS:
Overall Officials: Ali Alagoz, Assoc Prof, Principal Investigator — Atatürk Chest Diseases and Chest Surgery Training and Research Hospital
Locations (1):
- University of Health Sciences, Ankara Atatürk Chest Diseases and Thoracic Surgery Training and Research Hospital, Keçiören, Ankara, Turkey (Türkiye)